CLINICAL TRIAL: NCT04435743
Title: The Efficacy and Safety of Lenalidomide With or Without Rituximab and Other Drugs in B-cell Non-Hodgkin Lymphomas: a Real-world Study.
Brief Title: Efficacy and Safety of Lenalidomide With or Without Rituximab and Other Drugs in B-cell Non-Hodgkin's Lymphomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director of Shanghai Institute of Hematology, Ruijin Hospital
Other Study IDs: LEN-NHL
Record Dates: First submitted 2020-05-20; First posted 2020-06-17 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Non-hodgkin Lymphoma,B Cell
Keywords: lenalidomide; Non-hodgkin Lymphoma,B Cell
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DLBCL: Treatment-naive or relapsed/refractory CD20+ diffuse large B-cell lymphoma patients who receive induction therapy containing lenalidomide.
  Interventions: Drug: Lenalidomide
- FL/MCL/MZL: Treatment-naive or relapsed/refractory CD20+ follicular lymphoma, mantle cell lymphoma and marginal zone lymphoma patients who receive induction therapy containing lenalidomide.
  Interventions: Drug: Lenalidomide
- Maintenance: B-cell non-Hodgkin lymphoma patients who achieve complete or partial remission after induction therapy and receive maintenance therapy containing lenalidomide.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide is given as any following dosage:
  1. 25mg, PO QD, Day 1-10 in every 21 days for 6 cycles;
  2. 15mg, PO QD, Day 1-14 in every 21 days for 6 cycles;
  3. 25mg, PO QD, Day 1-10 in every 21 days for 1 year;
  4. 25mg, PO QD, Day 1-21 in every 28 days for 1 year;
  5. 25mg, PO QD, Day 1-10 in every 28 days for 12 cycles;
  6. 20mg, PO QD, Day 1-21 in every 28 days for 12 cycles.

SUMMARY:
Describe the treatment of B-cell non-Hodgkin lymphoma patients who receive lenalidomide single drug or lenalidomide combined with rituximab (with or without other drugs), and evaluate the efficacy and safety of lenalidomide single drug or lenalidomide combined with rituximab (with or without other drugs) in the real-world setting.

DETAILED DESCRIPTION:
This is a multi-center prospective, observational real-world study, targeting patients with B-cell non-Hodgkin's lymphomas. This study is designed to evaluate the efficacy and safety of lenalidomide single drug or lenalidomide combined with rituximab (with or without other drugs) in the real-world setting.

This study will mainly focus on the following three cohorts:

Cohort 1: patients diagnosed with CD20-positive diffuse large B-cell lymphoma; Cohort 2: patients diagnosed with CD20-positive follicle lymphoma; Cohort 3: patients on maintenance treatment who have achieved complete remission or partial remission after induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as B-cell non-Hodgkin's lymphoma
* Voluntary participation in this study and the signing of an informed consent form
* The researchers assessed that the patient will benefit from the treatment of lenalidomide single drug or lenalidomide combined with rituximab (with or without other drugs)

Exclusion Criteria:

* Contradictions to any drug in the treatment regimen
* Pregnant or lactating women
* Patients who were not considered suitable for the study by the researchers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study focus on patients diagnosed with B-cell non-Hodgkin's lymphoma and treated with lenalidomide single drug or lenalidomide combined with rituximab (with or without other drugs) in the real-world setting.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | At the end of Cycle 6 (each cycle is 21-28 days)
  Rate of objective response, defined according to Lugano 2014 criterion.

SECONDARY OUTCOMES:
Complete response rate | At the end of Cycle 6 (each cycle is 21-28 days)
  Rate of complete response, defined according to Lugano 2014 criterion
Partial response rate | At the end of Cycle 6 (each cycle is 21-28 days)
  Rate of partial response, defined according to Lugano 2014 criterion
Duration of response | From response evaluation to study completion, an average of 2 years.
  Time to relapse or progression, measured from documentation of response, in CR or PR patients
2-year progression-free survival | 2 years after entry onto study
  The rate of patients who are free of disease progression or death as a result of any cause, measured from entry onto study, in all patients
Overall survival | From entry onto study to study completion, an average of 2 years.
  Death as a result of any cause, measured from entry onto study, in all patients
Adverse event | From entry onto study to study completion, an average of 2 years.
  any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure
Severe adverse event | From entry onto study to study completion, an average of 2 years.
  An adverse event when the patient outcome is death, life-threatening, required intervention to prevent permanent impairment or damage, hospitalization, disability or permanent damage, congenital anomaly or birth defect, or other important medical events
Dosage adjustment | From entry onto study to study completion, an average of 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China